CLINICAL TRIAL: NCT03761420
Title: Adjuvant Endocrine Therapy in Early Stage Breast Cancer: Impact of Drug Adherence/Persistence on Clinical Outcome in Various Breast Cancer Subtypes
Brief Title: Adjuvant Endocrine Therapy in Early Stage Breast Cancer: Adherence and Clinical Outcome
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/1356
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasm
Keywords: Medication Adherence; Antineoplastic Agents, Hormonal; Chemotherapy, Adjuvant; Treatment Outcome
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breast cancer postoperative: got surgery for breast cancer in St Olavs Hospital, Trondheim, during 2004-2013

SUMMARY:
Breast cancer is the most common cancer among women in Norway. In 2016, 3402 new cases were diagnosed (3371 in women). Breast cancer is still the second most common cause of death from cancer among women with 585 breast cancer deaths in Norway in 2015. The majority of the patients (70-75 %) belong to the Luminal subtypes, which comprise the hormone receptor (oestrogen receptor (ER) and/or progesterone receptor (PR)) positive tumours.

The most important systemic adjuvant therapy in luminal breast cancers is a long-lasting administration of per-oral anti-oestrogen medication. A systemic hypo estrogenic state in the body may be created by the selective oestrogen receptor modulator tamoxifen or by inhibitors of the peripheral systemic aromatization of adrenal androgens into estrogens (aromatase inhibitors). Initially, tamoxifen was given adjuvant for 2 years, later prolonged to 5 years and recently an extension to 10 years has been recommended for premenopausal women. Aromatase inhibitors were introduced in Norwegian treatment guidelines in 2002. Currently, they are recommended in postmenopausal patients for 5 years, either as monotherapy or in concert with tamoxifen (aromatase inhibitors for 2 years followed by tamoxifen for 3 years).

In premenopausal breast cancer patients, tamoxifen still is the drug of choice. Two of the major underlying reasons for late recurrences in luminal breast cancer subtypes are development of endocrine resistance to tamoxifen and aromatase inhibitors or failure of taking the medication as prescribed. Higher mortality has been shown for breast cancer patients with reduced tamoxifen adherence. The patients' ability to follow instructions and recommendations are probably overestimated in controlled trials due to patient selection and close follow-up in the study setting. Some patients experience distressing side effects like hot flushes, fatigue, joint pain, mood swings and vaginal dryness. To the investigators' knowledge, there are few studies in Norway regarding discontinuation of endocrine treatment in breast cancer. In this study they will investigate the long-term discontinuation pattern to oral adjuvant systemic endocrine therapy in a large cohort of breast cancer patients treated in St. Olav's hospital in Trondheim, Norway, and the association between adherence to endocrine treatment and long-term survival.

DETAILED DESCRIPTION:
After identifying all patients who were recommended endocrine therapy, data will be linked to the Norwegian Prescription Database (NorPD). Adherence will be estimated based on to which extent the patients actually have effectuated their prescriptions at Norwegian pharmacies. In the 5-year long treatment period, the patients receive a prescription refill of tamoxifen or aromatase inhibitor tablets for a 100 days interval. Medication Possession Ratio (MPR) will be used as proxy for adherence. The estimations will be performed in the following way: For each patient, we will receive the total number of pills and the total length of time from first to latest prescription effectuated. MPR is the number of pills divided by the total number of days in the time from first prescription to discontinuation. Discontinuation will be estimated to date for latest effectuation of the prescription plus 100 days (due to the number of pills prescribed). From these estimations, we will categorize the patients in groups taking MPR and total period of time into consideration. Taking prescript medication equal to or more than 80% is considered as adherent (MPR ≥ 80 %). Likewise, non-adherence is defined as MPR < 80 %.

ELIGIBILITY:
Inclusion Criteria:

Luminal breast cancer

Exclusion Criteria:

Non-Luminal breast cancer

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients treated (surgery) at St Olavs Hospital in Trondheim, Norway, during 2004-2013.
Sampling Method: Non-Probability Sample
Enrollment: 1411 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio (MPR) as a proxy for medication adherence | 0-5 years after surgery for breast cancer
  see Detailed description
Survival | 5-14 years after surgery for breast cancer
  Breast cancer specific survival according to adherence and non-adherence

CONTACTS AND LOCATIONS:
Overall Officials: Anne Irene Hagen, md phd, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway